CLINICAL TRIAL: NCT05705310
Title: The STRENGTH Study: Self-management and Theory-based Rehabilitation Encouraging New Gateways to Healthy-Hearts
Brief Title: Self-management and Theory-based Rehabilitation Encouraging New Gateways to Healthy-Hearts
Acronym: STRENGTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health Development Unit (Unknown); Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RG3_20-1-3.Z
Record Dates: First submitted 2023-01-06; First posted 2023-01-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-02

CONDITIONS: Coronary Disease
Keywords: Cardiac rehabilitation; Exercise; Secondary prevention
MeSH Terms: conditions — Coronary Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomised controlled trial design will be employed involving random and sequential crossover of clusters from control to intervention until all clusters are exposed
Who Masked: Outcomes Assessor
Masking Description: A separate researcher, not involved in the delivery of the intervention or assessment of outcomes, will generate the randomisation sequence which will be concealed in sealed opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Self Management Strategies
- Control Group (No Intervention): Individuals in the control group will receive usual care

INTERVENTIONS:
Behavioral: Self Management Strategies — During their maintenance stage cardiac rehabilitation programme, participants will be given a pedometer and asked to wear it during waking hours to record their daily step counts and/or time in physical activity each week. Participants will be encouraged to gradually achieve 150 minutes of moderate-intensity exercise per week and self-monitor their progress using the pedometer. At the end of every week, participants will review progress and set goals with an exercise professional. Group discussions will also take place, focusing on the benefits of regular physical activity, demonstrating lifestyle activities that can help accumulate activity and identifying various means of social support, and identifying local opportunities (groups or places) for physical activity after the cardiac rehabilitation programme has ended. Following this, they will receive a monthly phone call from the exercise professional to check progress and encourage them to continue with the programme.
  Arms: Intervention Group

SUMMARY:
The goal of this intervention is translate current behaviour change in to community cardiac rehabilitation programmes for people living beyond a heart attack. The main question it aims to answer is whether adding a lifestyle change programme promoted maintenance of physical activity changes will be maintained following a cardiac rehabilitation programme.

The problem Guidelines recommend that coronary heart disease patients should be offered cardiac rehabilitation which includes exercise programmes, education, and ongoing support within both clinical and community settings. Cardiac rehabilitation programmes reduce the risk of death and illness, but it is likely that patients will stop exercising without enough support. New was to encourage coronary heart disease patients to stay active both during and after taking part in cardiac rehabilitation programmes are needed.

The project Behaviour change techniques can encourage patients to stay active for longer. The aim of this project is to see whether behaviour change can encourage coronary heart disease patients taking part in community-based cardiac rehabilitation programmes to stay active for longer compared with patients receiving the standard cardiac rehabilitation programme.

The benefits It is hoped that these methods will encourage more cardiac rehabilitation patients to stay physically active for longer and improve health. The results will provide more evidence on using behavioural change techniques in cardiac rehabilitation programmes and have the potential to benefit many patients with coronary heart disease throughout Northern Ireland and the rest of the United Kingdom.

DETAILED DESCRIPTION:
Coronary heart disease is the leading cause of death and disability worldwide. Guidelines recommend that all coronary heart disease patients should be offered cardiac rehabilitation which includes exercise programmes, education, and ongoing support within both clinical and community settings following a heart-related event, surgery or procedure.

The core cardiac rehabilitation programme (previously known as Phase III) is delivered by a clinical team in hospital. Depending on the location, it may involve a combination of exercise training, health education, and advice on reducing the risk of having a heart-related event such as ways to manage stress. After the patients complete this programme, participants are assessed for suitability to attend a community-based exercise programme called the maintenance cardiac rehabilitation programme (previously Phase IV). Cardiac rehabilitation programmes reduce the risk of death and illness, but evidence shows that it is unlikely that patients will maintain the required exercise levels without the support and structure provided by such exercise programmes. A previous study found that using behaviour change techniques, such as problem-solving skills, encouraged participants to stay active for longer. New ways to encourage coronary heart disease patients to stay active both during and after taking part in cardiac rehabilitation programmes are needed. The aim of this project is to translate behaviour change research in a cardiac rehabilitation programme to encourage coronary heart disease patients to stay active for longer.

The aim of this project is to translate behaviour change research into current maintenance stage (Phase IV) cardiac rehabilitation services. The hypothesis is that by adding a lifestyle change programme promoting self-efficacy, physical activity (PA) changes will be maintained following a cardiac rehabilitation programme.

All participants will be recruited while taking part in Active Belfast maintenance stage cardiac rehabilitation (CR) programmes. Participants will have already completed the Phase III core cardiac rehabilitation programme and been assessed for suitability to take part in the study. Some participants will be randomly chosen to receive the intervention which includes additional sessions to encourage active lifestyles. This will involve wearing a pedometer to count steps. Each week, participants will report their step counts and review their goals. In week eight, participants will have a group discussion with the researcher during which participants will discuss the benefits of physical activity. In week twelve, there will be a second group discussion about potential barriers to being active with advice on practical ways to do more activity. Participants will receive a monthly phone call from the exercise professional to check their progress and encourage them to adhere to the programme and achieve their weekly goals.

Participants in the control group will receive the standard cardiac rehabilitation maintenance programme. After the study, all participants will receive a pedometer and be given instructions on how to use it as well as a booklet from the Public Health Agency to advise them on how to increase their physical activity. Participants' physical activity will be measured using activity monitors at the beginning of the study, at twelve weeks (end of maintenance stage cardiac rehabilitation programme) and then at six months. Body measurements such as height, weight and blood pressure will also be taken, as well as a measure their physical and mental health. The difference in steps and time spent in moderate-vigorous physical activity between the intervention group and the control group after six months will be analysed. How well the intervention has been completed by participants (i.e. attendance records) and delivered by the exercise professional (i.e. satisfaction with the programme) will be assessed through interviews and focus groups. The cost-effective the study will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participants referred to a maintenance stage cardiac rehabilitation programme

Exclusion Criteria:

* Individuals who do not wish to provide consent to participate in this study or cannot commit to the full 12 weeks of the CR programme will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Steps per Day in the last seven days | Change from baseline steps per day at 6 months
  Measured using a validated ActiGraph GT3X+ accelerometer worn for 7 consecutive days
Time spent in moderate-vigorous intensity physical activity in the last seven days | Change from baseline time spent in moderate-vigorous intensity physical activity at 6 months
  Measured using a validated ActiGraph GT3X+ accelerometer worn for 7 consecutive days

SECONDARY OUTCOMES:
Physical activity self efficacy | Change from baseline physical activity self-efficacy at 6 months
  Physical activity self-efficacy scale. This scale includes nine items, each rated on a scale from 1 to 10. The minimum possible score is 9 and maximum score is 90, with higher scores indicating better self-efficacy.
Physical and mental health | Change from baseline physical and mental health at 6 months
  Measured using the self reported Short-form 12 (SF-12) Health Survey questionnaire
Mental wellbeing | Change from baseline mental wellbeing at 6 months
  Measured using the self reported Warwick-Edinburgh Mental Well-being Scale (WEMWBS). This scale includes 14 items, each rated on a scale from 1 to 5. The minimum possible score is 14 and maximum score is 70, with higher scores indicating better metal wellbeing.
Health-related quality of life | Change from baseline quality of life at 6 months
  Measured using the self reported EuroQol-5D-3L questionnaire
Blood pressure | Change from baseline systolic and diastolic blood pressure at 6 months
  Resting systolic and diastolic blood pressure measured using a digital sphygmomanometer
Body mass index | Change from baseline body mass index at 6 months
  Body mass divided by the square of height
Waist and hip circumference | Change from baseline waist and hip circumference at 6 months
  Waist circumference will be measured as the midpoint between the lowest rib and the iliac crest, using a fibre glass tape.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole E Blackburn, PhD, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.